CLINICAL TRIAL: NCT04758208
Title: Establishment of Pediatric Reference Intervals for Mindray Hematology Parameters for Worldwide Application in Clinical Laboratories
Brief Title: Mindray Pediatric Hematology Reference Intervals Study
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: MINDRAY (Unknown)
Responsible Party: Principal Investigator, Khosrow Adeli, Head of Clinical Biochemistry, The Hospital for Sick Children
Other Study IDs: REB1000069402
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Establish Hematology Reference Intervals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Fresh whole blood specimens will be collected in K2EDTA tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy CALIPER Participants: Healthy community children and adolescents recruited through the CALIPER initiative as well as healthy children and adolescents recruited from outpatient clinics at the Hospital for Sick Children through the CALIPER initiative. Blood samples from these participants will be tested on the Mindray BC-6800Plus device to measure hematology parameters and establish reference intervals.
  Interventions: Diagnostic Test: Hematology Parameters

INTERVENTIONS:
Diagnostic Test: Hematology Parameters — Measurement of hematology parameters on BC-6800Plus

SUMMARY:
This study is a collaborative initiative between the CALIPER (Canadian Laboratory Initiative on Pediatric Reference Intervals) program at the Hospital for Sick Children (HSC) and Mindray Medical International Limited to establish a database of pediatric reference intervals for hematology parameters on BC-6800Plus.

DETAILED DESCRIPTION:
The purpose of this study is to establish accurate and robust ethnic-, age- and sex-specific reference intervals for hematology parameters during childhood and adolescence on the Mindray analyzer (BC-6800Plus).

Subjects will be recruited for this study through the CALIPER initiative and will include healthy children and adolescents in the community and in outpatient clinics at the Hospital for Sick Children (HSC). Since all participants will be recruited through the CALIPER initiative, the CALIPER consent forms will be used to obtain consent from each child and their parent/guardian. These forms obtain consent to use the samples to develop reference intervals for a range of tests. This study aims to measure hematology parameters in these samples and is therefore encompassed within the CALIPER consent. Recruitment will focus on subjects from three ethnic groups: Caucasians, Hispanics, and South Asians. A total of 960 subjects will be recruited for this study through the CALIPER initiative. The total sample size was determined by considering the requirement of 60-120 samples per partition for five age groups (0-<1 years, 1-<5 years, 5-<10 years, 10-<15 years, 15-<19 years). Each age group will consist of an equal number of females and males. Additional samples may be required if data analysis suggests further age and/or sex partitioning for specific parameters.

Each subject will provide a blood sample, which will be collected through the CALIPER initiative. These samples will be analyzed as part of this study in a secondary-use/retrospective fashion. Specifically, fresh whole blood specimens will be collected in K2EDTA tubes, placed in biohazard bags, stored on ice, and analyzed on the Mindray hematology platform within 8 hours of collection. All available hematology parameters for the BC-6800Plus will be measured (37 report and 48 research hematology parameters, as per the user manual). All procedures will be performed according to the user manual. Mindray quality control materials will be used to monitor the performance of the assays during the study. HSC will retain all quality controls data, maintenance record and reagents/calibrators lot numbers. Quality controls will be run daily and analysis of the CALIPER samples will proceed only after all the quality control (QC) data are acceptable.

Data analysis will be performed by the CALIPER team in accordance with Clinical & Laboratory Standards Institute (CLSI) EP28-A3c guidelines on defining, establishing, and verifying reference intervals in the clinical laboratory. The statistical approach for reference interval establishment has been described in-depth previously. In brief, analyte concentrations will be plotted against age and colour-coded by sex. Following visual inspection, extreme outliers will be removed and suspected age- and sex-specific partitions will be confirmed using the Harris and Boyd statistical method. Normality of data will be qualitatively assessed using quantile-quantile plots and quantitatively assessed using the Shapiro-Wilk's test. If skewed, the Box-Cox transformation will be applied in an effort to transform the data to a normal distribution. Outliers will be subsequently identified and removed using the Tukey or adjusted Tukey method for Gaussian and non-Gaussian data distributions, respectively. Reference intervals for partitions with ≥120 participants will be calculated using the nonparametric method. Reference intervals for partitions with ≥40 and <120 participants (60 for group 0-<1 years and 1-<5 years, 120 for group 5-<10 years, 10-<15 years and 15-<19 years) will be calculated using the robust method. 90% percent confidence intervals will also be calculated for the lower and upper limit of each reference interval. Ethnic-specific reference intervals will be calculated if sample size for each ethnic group is adequate. Otherwise, reference value distributions for South Asian and Hispanic children will be compared to those of Caucasian children.

Oversight Authority (additional information)

* This study is regulated by 'Canada: Health Canada'
* This study has been reviewed and approved by 'Canada: Ethics Review Committee'

ELIGIBILITY:
Inclusion Criteria:

* 0-<19 years

Exclusion Criteria:

* History of chronic illness
* Use of prescription medications within 2 weeks of collection
* Acute illness within 7 days of collection
* Pregnancy

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy community children and adolescents as well as healthy children and adolescents recruited from outpatient clinics at the Hospital for Sick Children.
Sampling Method: Non-Probability Sample
Enrollment: 691 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
White Blood Cell count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Basophil number | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Basophil percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Neutrophil number | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Neutrophil percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Eosinophil number | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Eosinophil percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Lymphocyte number | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Lymphocyte percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Monocyte number | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Monocyte percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Immature Granulocyte number | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Immature Granulocyte percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Reticulocyte percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Reticulocyte number | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Reticulocyte Hemoglobin Expression | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Immature reticulocyte fraction | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Low fluorescent ratio | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Middle fluorescent ratio | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
High fluorescent ratio | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Red blood cell count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Hemoglobin Concentration | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Mean Corpuscular Volume | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Mean Corpuscular Hemoglobin | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Mean Corpuscular Hemoglobin Concentration | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Red Blood Cell Distribution Width - Coefficient of Variation | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Red Blood Cell Distribution Width - Standard Deviation | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Hematocrit | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Nucleated red blood cell (NRBC) number | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Nucleated red blood cell percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Platelet count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Mean Platelet Volume | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Platelet Distribution Width | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Plateletcrit | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Immature Platelet Fraction | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Platelet-large cell ratio | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Platelet-large cell count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer

SECONDARY OUTCOMES:
High fluorescent Cell number | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
High fluorescent Cell percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Optical Red Blood Cell count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Optical Platelet count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Platelet count - Impedance | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Optical White Blood Cell count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
White blood cell counts - Differential (DIFF) | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Total nucleated cell counts - DIFF | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Immature Eosinophil percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Immature Eosinophil number | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
High forward scatter NRBC ratio | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Low forward scatter NRBC ratio | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Neutrophil-to-lymphocyte ratio | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Platelet-to-lymphocyte ratio | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
White blood cell count - white cell nucleated basophil channel (WNB) | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Total nucleated cell counts | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Infected Red Blood Cell count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Infected Red Blood Cell permillage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Microcyte count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Microcyte percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Macrocyte count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Macrocyte percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Mean Reticulocyte Volume | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Red Blood Cell Fragment Count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Red Blood Cell Fragment Percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Platelet Distribution Width Standard Deviation | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Reticulocyte Production Index | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
High fluorescent Immature Platelet Fraction | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Immature Platelet Count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
DIFF scattergram, mean neutrophil distribution-side scatter intensity | Within 8 hours of sample collection
  Scattergram of laboratory values derived from the Mindray BC-6800Plus Auto Hematology Analyzer
DIFF scattergram, mean neutrophil distribution-side fluorescent light intensity | Within 8 hours of sample collection
  Scattergram of laboratory values derived from the Mindray BC-6800Plus Auto Hematology Analyzer
DIFF scattergram, mean neutrophil distribution-forward scatter intensity | Within 8 hours of sample collection
  Scattergram of laboratory values derived from the Mindray BC-6800Plus Auto Hematology Analyzer
DIFF scattergram, mean lymphocyte distribution-side scatter intensity | Within 8 hours of sample collection
  Scattergram of laboratory values derived from the Mindray BC-6800Plus Auto Hematology Analyzer
DIFF scattergram, mean lymphocyte distribution-side fluorescent intensity | Within 8 hours of sample collection
  Scattergram of laboratory values derived from the Mindray BC-6800Plus Auto Hematology Analyzer
DIFF scattergram, mean lymphocyte distribution-forward scatter intensity | Within 8 hours of sample collection
  Scattergram of laboratory values derived from the Mindray BC-6800Plus Auto Hematology Analyzer
DIFF scattergram, mean monocyte distribution-side scatter intensity | Within 8 hours of sample collection
  Scattergram of laboratory values derived from the Mindray BC-6800Plus Auto Hematology Analyzer
DIFF scattergram, mean monocyte distribution-side fluorescent light intensity | Within 8 hours of sample collection
  Scattergram of laboratory values derived from the Mindray BC-6800Plus Auto Hematology Analyzer
DIFF scattergram, mean monocyte distribution-forward scatter intensity | Within 8 hours of sample collection
  Scattergram of laboratory values derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Dimorphic population, smaller distribution RBC count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Dimorphic population, larger distribution RBC count | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Dimorphic population, smaller distribution mean corpuscular volume | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Dimorphic population, larger distribution mean corpuscular volume | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Mean Corpuscular Hemoglobin of Reticulocyte | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Mean Hemoglobin Distribution Width of Red Blood Cell | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Mean Platelet Concentration | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Mean Platelet Matter Content | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Hyperchromic Red Blood Cell percentage (Hyper%) | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer
Hypochromic Red Blood Cell percentage | Within 8 hours of sample collection
  Laboratory value derived from the Mindray BC-6800Plus Auto Hematology Analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Khosrow Khosrow, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Summary collated and anonymized data for each test available on the BC-6800Plus platform will be presented in the form of:
  * Scatter plots of anonymized test results plotted by age and colour-coded by sex.
  * Tables of established reference intervals, partitioned by age, sex, and ethnicity, if applicable.
  To ensure that the knowledge gained from this study will be disseminated and available to all pediatric healthcare centres, laboratories, and pediatrician offices, our knowledge translation strategies include:
  * Submission of data for publication to a peer-reviewed journal.
  * Full data will be made available electronically via an online secure database on the CALIPER website and mobile app to facilitate access for the pediatric healthcare community internationally.